CLINICAL TRIAL: NCT02513667
Title: Phase II Trial of Ceritinib in Combination With Stereotactic Ablative Radiation in ALK-rearranged Metastatic Lung Adenocarcinoma
Brief Title: Ceritinib in Combination With Stereotactic Ablative Radiation Metastatic Lung Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after UTSW was informed by Novartis that further support for the study would not be provided
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sawsan Rashdan, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 042015-076
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2021-12-17 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: ALK-positive Non-small Cell Lung Cancer
MeSH Terms: interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALK-inhibitor naive patients (Experimental): Patients will receive ceritinib at a dose of 750 mg (150 mg capsules times 5 capsules once a day) for 10 weeks. Patient will stop taking Ceritinib 72 hours before SABR (Stereotactic ablative body radiation). They could get 1, 3 ,or 5 treatments on consecutive days with 18 hours between each treatment or every other day (doctor's determination). The patient may start taking Ceritinib again 72 hours after radiation is complete. Patient will continue to take certinib for up to 8 months. At Follow-Up treatment, patients will be contacted every 3 months for 9 months.
  Interventions: Drug: Ceritinib; Radiation: Stereotactic ablative body radiation
- Patients recieved prior ALK inhibitor (Experimental): Patients will receive ceritinib at a dose of 750 mg (150 mg capsules times 5 capsules once a day) for 10 weeks. Patient will stop taking Ceritinib 72 hours before SABR (Stereotactic ablative body radiation). They could get 1, 3 ,or 5 treatments on consecutive days with 18 hours between each treatment or every other day (doctor's determination). The patient may start taking Ceritinib again 72 hours after radiation is complete. Patient will continue to take certinib for up to 8 months. At Follow-Up treatment, patients will be contacted every 3 months for 9 months.
  Interventions: Drug: Ceritinib; Radiation: Stereotactic ablative body radiation

INTERVENTIONS:
Drug: Ceritinib — Patients will receive ceritinib at a dose of 750 mg (150 mg capsules times 5 capsules once a day) for 10 weeks. Patient will stop taking Ceritinib 72 hours before SABR radiation. The patient may start taking Ceritinib again 72 hours after radiation is complete. Patient will continue to take certinib for up to 8 months.
Radiation: Stereotactic ablative body radiation — Patients will receive study drug for 10 weeks. They could get 1, 3 ,or 5 treatments on consecutive days with 18 hours between each treatment or every other day (doctor's determination).

SUMMARY:
The purpose of this study is to see if Ceritinib can target ALK in non-small cell lung cancer and slow down cancer growth and prevent it from spreading.

DETAILED DESCRIPTION:
This is an, open-label, two-cohort protocol designed to evaluate the activity of targeted therapy and SABR in ALK positive lung adenocarcinoma.

Cohort A will evaluate the combination in ALK-inhibitor naïve patients. Cohort B will evaluate the combination in patients who have received treatment with one prior ALK inhibitor.

Ceritinib will be administered to the patient until disease progression by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or discontinuation of the trial for any other reason including death.

The primary focus of this protocol is identifying response in ALK+ lung cancer patients. Patients with Ventana assay and Vysis FISH probe positive tumors will be treated. Evidence of ALK gene rearrangement will also be considered eligible for the trial.

Primary Objective:

Cohort A: Superiority of ceritinib + SABR median PFS compared to historical control of 10 months (expected to be 20 months)

Endpoint:

Cohort A Median PFS defined as time from initiation of ceritinib until disease progression by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or discontinuation of the trial for any other reason including death.

Primary:

Cohort B: Superiority of ceritinib + SABR median PFS compared to historical control of 7 months.

Endpoint:

Cohort B: Median PFS defined as time from initiation of ceritinib until disease progression by RECIST 1.1, unacceptable toxicity, withdrawal of consent, or discontinuation of the trial for any other reason including death.

Secondary:

* Report Overall survival Overall survival
* Report Time to 2nd SABR Time from start of systemic therapy to first day of second course of SABR
* Report Time to 3rd SABR Time from start of therapy to first day of third course of SABR
* Report proportion of patients CR/PR/stable disease at 6 and12 months Number of patients with CR/PR/stable disease for 6 and 12 months after initiation

Safety:

-Demonstrate safety of ceritinib followed by SABR Describe toxicity and adverse events (CTCAE v.4) compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of lung adenocarcinoma that demonstrates ALK rearrangement as detected by the approved FISH test (Abbott Molecular Inc), using Vysis breakapart probes (defined as 15% or more positive tumor cells); or the Ventana IHC test. Evidence of rearrangement by gene sequencing tests such as FoundationOne or Caris will also be seen as evidence of ALK abnormality and meeting eligibility requirement.
2. Patients with no prior ALK-inhibitor therapy will be placed in cohort A, those treated with one prior line of ALK-inhibitor (at any time) will enter cohort B.
3. Patients will not have any other curative therapeutic option, such as radiation or surgery.
4. WHO performance status 0-2.
5. Age ≥18 years.
6. Patients must have recovered from all toxicities related to any prior anticancer therapies to ≤ Grade 2 (CTCAE v 4.03), provided that any concomitant medication is given prior to initiation of treatment with ceritinib. Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.
7. Adequate organ function: the following laboratory criteria have been met:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin (Hgb) ≥ 8 g/dL
   * Platelets ≥ 75 x 109/L
   * Serum creatinine <1.5 mg/dL and /or calculated creatinine clearance (using Cockcroft-Gault formula) ≥30 mL/min
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN), except for patients with Gilbert's syndrome who may be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
   * Aspartate transaminase (AST) < 2.0 x ULN, except for patients with liver metastasis, who are only included if AST < 3 x ULN; alanine transaminase (ALT) < 2.0 x ULN, except for patients with liver metastasis, who are only included if ALT < 3 x ULN
   * Alkaline phosphatase (ALP) ≤5.0 x ULN
   * Fasting plasma glucose ≤175 mg/dL (≤9.8 mmol/L)
   * Serum amylase ≤ 2 x ULN
   * Serum lipase ≤ ULN
8. Patient must have the following laboratory values or have the following laboratory values corrected with supplements to be within normal limits before the first dose of ceritinib:

   * Potassium
   * Magnesium
   * Phosphorus
   * Total calcium (corrected for serum albumin)
9. Written informed consent for the protocol must be obtained prior to any screening procedures.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

1. Patients with known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate).
2. History of carcinomatous meningitis.
3. Prior therapy with ceritinib.
4. Presence or history of a malignant disease other than lung adenocarcinoma that has been diagnosed and/or required therapy within the past year and is undergoing active anticancer treatment. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
5. Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
6. Patient who has received thoracic radiotherapy to lung fields ≤4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs) radiotherapy ≤2 weeks prior to starting the study treatment or has not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤2 weeks prior to starting study treatment is allowed.
7. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

   * unstable angina within 6 months prior to screening;
   * myocardial infarction within 6 months prior to screening;
   * history of documented congestive heart failure (New York Heart Association functional classification III-IV);
   * uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication
   * initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
   * ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication;
   * other cardiac arrhythmia not controlled with medication;
   * Corrected QT (QTcF) >470 ms using Fridericia's correction on the screening ECG
8. Impaired GI function or GI disease that may alter absorption of ceritinib or inability to swallow up to five ceritinib capsules daily. Although, patients unable to swallow capsules will be allowed to participate in this study, by following the specific instructions on making a slurry of the medication.
9. Patient has impairment of GI function or GI disease that may significantly alter the absorption of ceritinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
10. Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with ceritinib and for the duration of participation (see Appendix 1 Tables):

    * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
    * Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, CYP2C8 and/or CYP2C9 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (eg, dabigatran, rivaroxaban, apixaban).
    * Unstable or increasing doses of corticosteroids; If patients are on corticosteroids for endocrine deficiencies or tumor-associated symptoms (non-CNS), dose must have been stabilized (or decreasing) for at least 5 days before first dose of study treatment.
    * Enzyme-inducing anticonvulsive agents
    * Herbal supplements
11. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and agree to continue for 3 months after the last dose of study treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of any two of the following (a+b or a+c or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

    In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
13. Sexually active males unless they agree to use a condom during intercourse while taking drug and agree to continue for 3 months after the last dose of study treatment. Male patients for 3 months should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
14. Patient has a history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.
15. Patient has other severe, acute, or chronic medical conditions including uncontrolled diabetes mellitus or psychiatric conditions or laboratory abnormalities that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
16. Patient has had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior to starting study treatment or has not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can receive study treatment ≥1 week after these procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2021-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Khan, MD, Principal Investigator — UT Southwetern Medical Center-Oncology
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Started | 8 | 6
Completed | 8 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 patient withdrew consent before thier first scan.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Number of days until disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Baseline until date of first observed disease progression or death, assessed up to 31.7 months.
Measure: Mean (Full Range); unit: days
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 8 | 5
days | 505 [350 to 747] | 482 [73 to 963]

2. Secondary Outcome: Overall Survival
Description: Overall survival is the percentage of participants alive at the given time point. OS is defined as the time to death from the start of drug therapy.
Time Frame: at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 8 | 5
Participants | 8 | 5

3. Secondary Outcome: Time to 2nd Subsequent Stereotactic Ablative Radiation
Description: After the initial SABR to persisting lesions, if new lesions appear or if existing lesions enlarge but are amenable to SABR, patients will remain on study and listed as not having progressed. Time from start of systemic therapy to first day of second course of SABR
Time Frame: 18 hours
Population: No patients received a second course of SABR
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to 3rd Subsequent Stereotactic Ablative Radiation (SABR)
Description: Time from start of therapy to first day of third course of SABR was measured.
Time Frame: 3 months
Population: Data was not collected due to early termination of the study since no participant received 3rd SABR.
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Patients With CR/PR/Stable Disease for 6 Months
Description: Number of patients with CR/PR/stable disease for 6 months was measured by evaluating target lesions.
  Complete Response (CR): Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 8 | 5
Participants | 2 | 1

6. Secondary Outcome: Number of Patients With CR/PR/Stable Disease for 12 Months
Description: Number of patients with CR/PR/stable disease for 12 months was measured by evaluating target lesions.
  Complete Response (CR): Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 8 | 5
Participants | 2 | 2

7. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
Number analyzed (Participants) | 8 | 5
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: Baseline until date of first observed disease progression or death, an average of 12 months
Arm/Group | ALK-inhibitor Naive Patients | Patients Recieved Prior ALK Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/5
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALK-inhibitor Naive Patients (N=8) | Patients Recieved Prior ALK Inhibitor (N=5)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALK-inhibitor Naive Patients (N=8) | Patients Recieved Prior ALK Inhibitor (N=5)
Abdominal Pain (Gastrointestinal disorders) | 4 | 3
Acid Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (6) | 3 (5)
Increased ALT (Investigations) | 4 (7) | 2 (6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Appetite Change (dysgeusia, anorexia, decreased appetite) (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Increased AST (Investigations) | 3 (6) | 3 (3)
Pain - Back (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Benign Familial Tremmors (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 2 (2) | 2 (2)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Pain - BL Foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Burning sensation (General disorders) | 1 (2) | 1 (1)
Chest Pain (Cardiac disorders) | 3 (5) | 1 (2)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0)
cold (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Hypertnesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypercholesterolemia (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased Creatinine (Renal and urinary disorders) | 1 | 3 (5)
cough (General disorders) | 2 (2) | 3 (3)
intraoperative ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased ANC (General disorders) | 0 (0) | 1 (1)
Decreased calcium (General disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (9)
Impaired Balance (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Disequilibrium (Nervous system disorders) | 1 (1) | 0 (0)
Discomfort in the sciatic nerve right leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Discomfort left side of rib cage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Increased GGT (Investigations) | 2 (3) | 1 (3)
Increased Lipase (Investigations) | 1 (1) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Flu like symptoms (achy,warm) (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes Simplex (Immune system disorders) | 1 (1) | 0 (0)
Increased amylase (Investigations) | 1 (1) | 2 (4)
Increased blood bilirubin (Investigations) | 1 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Increased lymphocyte (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Vomitting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Intermittent bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pain- Knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Intermittent hand and finger spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash (Immune system disorders) | 2 (2) | 1 (1)
stomach cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Latent tuberculosis (General disorders) | 1 (1) | 0 (0)
Tooth Infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Low albumin (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malignant pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - right lung, shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right Leg/Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - General (General disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Prolonged QT (Investigations) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus (hands) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seasonal allergies (Immune system disorders) | 3 (3) | 1 (1)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infections: shingles (Infections and infestations) | 0 (0) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
T wave abnormality (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Vascular disorders) | 1 (1) | 0 (0)
Tranaminatis (General disorders) | 0 (0) | 1 (1)
Trapped Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Worsening Allergies (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02513667/Prot_SAP_000.pdf